CLINICAL TRIAL: NCT00257621
Title: A Pilot, Phase II, Open-label, Single Arm Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of GW640385 When Administered With Ritonavir in Combination With NRTIs for 48 Weeks in HIV-1 Infected Adults
Brief Title: GW640385 Plus Ritonavir And NRTIs For 48 Weeks In HIV-1 Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPR10006
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Infection, Human Immunodeficiency Virus I; HIV Infection
Keywords: HIV-1 protease inhibitor GW640385 ritonavir RTV
MeSH Terms: conditions — Infections; HIV Infections | interventions — Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW640385
Drug: Ritonavir
  Other Names: GW640385

SUMMARY:
This is a proof of concept (POC) single arm study of GW640385, a protease inhibitor, in combination with RTV and 2 or more nucleoside reverse transcriptase inhibitors (NRTI) backbone. This study has a 48 week duration and is open to both treatment naive and experienced patients who are HIV positive. There are 3 intensive pharmacokinetic (PK) visits.

ELIGIBILITY:
Inclusion criteria:

* HIV-1 infected subjects.
* Females must be of either non-childbearing potential or have a negative pregnancy test at Screening and agree to use a protocol approved method of contraception.
* Plasma HIV-1 RNA (viral load) >/=1,000 copies/mL at Screening.
* CD4+ cell count >/= 200 cells/mm3 at Screening.
* Be able to receive at least two of the following NRTIs (3TC, FTC, d4T, ddI or ZDV)to build a nucleoside backbone regimen.
* Willing and able to provide signed and dated written informed consent prior to study entry.

Exclusion criteria:

* Active CDC Class C disease.
* Pregnant or breastfeeding women.
* Protocol-specified laboratory abnormalities at Screening.
* Personal or family history of autoimmune disease.
* History or current indication of thyroid dysfunction or current thyroid gland abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with plasma HIV-1 RNA <400 copies/ml. Incidence of serious adverse events, rash and thyroid function abnormalities. GW640385 PK parameters. | throughout the study

SECONDARY OUTCOMES:
Changes over time in HIV-1 viral load and CD4+ cell counts. Incidence of adverse events and laboratory abnormalities. GW640385 and RTV PK parameters. Development of resistance in subjects with virologic failure. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (9):
- United States (9):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Seattle, Washington